CLINICAL TRIAL: NCT01629758
Title: A Phase 1 Dose Escalation Study of BMS-982470 (Recombinant Interleukin-21, rIL-21) in Combination With BMS-936558 (Anti-PD-1) in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: Safety Study of IL-21/Anti-PD-1 Combination in the Treatment of Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA220-008
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Neoplasms by Site
MeSH Terms: conditions — Neoplasms by Site | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1-Arm A: BMS-982470 (weekly x 4) + BMS-936558 (Experimental): Dose Escalation BMS-982470 10, 30, 50, 75 or 100 µg/kg Solution, Intravenous, During each 6 week cycle: weekly x 4 (i.e during weeks 1 through 4), Up to 2 years + BMS-936558 3 mg/kg Solution, Intravenous, During each 6 week cycle: every other week (i.e during weeks 1, 3, and 5), Up to 2 years
  Interventions: Biological: Denenicokin; Biological: Nivolumab
- Part 1-Arm B: BMS-982470 (3 times/week) + BMS-936558 (Experimental): Dose Escalation BMS-982470 10, 30, 50, 75 or 100 µg/kg Solution, Intravenous, During each 6 week cycle: 3 times/week during weeks 1 and 3, Up to 2 years + BMS-936558 3 mg/kg Solution, Intravenous, During each 6 week cycle: every other week (i.e during weeks 1, 3, and 5), Up to 2 years
  Interventions: Biological: Denenicokin; Biological: Nivolumab
- Part 2-Arm A: BMS-982470 (weekly x 4) + BMS-936558 (Experimental): Cohort Expansion BMS-982470 (dose selected in Part 1) Solution, Intravenous, During each 6 week cycle: weekly x 4 (i.e during weeks 1 through 4), Up to 2 years + BMS-936558 3 mg/kg Solution, Intravenous, During each 6 week cycle: every other week (i.e during weeks 1, 3, and 5), Up to 2 years
  Interventions: Biological: Denenicokin; Biological: Nivolumab

INTERVENTIONS:
Biological: Denenicokin
  Other Names: BMS-982470; rIL-21(recombinant interleukin 21)
Biological: Nivolumab
  Other Names: BMS-936558; Anti-PD-1 (Anti-Programmed-Death-1); MDX-1106

SUMMARY:
The purpose of this study is to determine whether the combination of the 2 drugs being investigated (IL-21 and anti-PD-1) is safe, and provide preliminary information on the clinical benefits of two different schedules of the combination.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* All subjects will have locally advanced or metastatic solid tumors
* For Part 2 (Cohort Expansion):

  * Tumor types will be restricted to clear cell renal cell carcinoma (ccRCC), non-small cell lung cancer (NSCLC), and melanoma
* At least 1 lesion with measurable disease
* Only subjects with tumor samples that are PD-L1 positive or negative are eligible

Exclusion Criteria:

* Uncontrolled central nervous system (CNS) or leptomeningeal metastasis
* Inadequate liver or kidney function
* History of autoimmune Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Safety, as measured by the rate of adverse events and serious adverse events | Approximately up to 4.5 years

SECONDARY OUTCOMES:
Efficacy as measured by tumor assessment (RECIST) | Week 6 of for the first 4 cycles, Week 6 of alternate cycle starting with cycle 6, End of Treatment (2 years) and approximately every 12 weeks during follow-up (approximately 1 year)
  Based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 using Best overall response (BOR), Objective response rate (ORR), Duration of Response (DOR), Progression-Free Survival Rate (PFSR)
Immunogenicity as measured by incidence of specific antidrug antibodies (ADA) to BMS-98470 and BMS-936558 | Up to 2 years + 100 days post-treatment follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- United States (5):
  - Oncology Research Associates, Pllc D/B/A, Scottsdale, Arizona
  - Yale University School Of Medicine, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Sidney Kimmel Comprehensive Cancer Center At Johns Hopkins, Baltimore, Maryland
  - Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx